CLINICAL TRIAL: NCT07033026
Title: A Phase 2, Multicenter, Randomized, Double Blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of NGM120 in Participants With Colorectal Cancer Who Have Cancer Cachexia
Brief Title: An Evaluation of NGM120 in a Randomized, Double-blind, Placebo-controlled Study in Participants With Colorectal Cancer Who Have Cancer Cachexia.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120-CX-202
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; CRC (Colorectal Cancer); Cancer Cachexia
Keywords: Cancer Cachexia; Colorectal Cancer; CRC
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- NGM120 Treatment Group A (Experimental): NGM120 low dose given subcutaneously every 4 weeks
  Interventions: Drug: NGM120 Q4W
- NGM120 Treatment Group B (Placebo Comparator): Placebo low dose given subcutaneously every 4 weeks
  Interventions: Drug: Placebo given
- NGM120 Treatment Group C (Experimental): NGM120 high dose given subcutaneously every 4 weeks
  Interventions: Drug: NGM120 Q4W
- NGM120 Treatment Group D (Experimental): NGM120 high dose given subcutaneously every 8 weeks
  Interventions: Drug: NGM120 Q8W
- NGM120 Treatment Group E (Placebo Comparator): Placebo high dose given subcutaneously every 4 weeks
  Interventions: Drug: Placebo given

INTERVENTIONS:
Drug: NGM120 Q4W — NGM120 given subcutaneously every 4 weeks
  Arms: NGM120 Treatment Group A; NGM120 Treatment Group C
Drug: NGM120 Q8W — NGM120 given subcutaneously every 8 weeks
  Arms: NGM120 Treatment Group D
Drug: Placebo given — Placebo given subcutaneously every 4 weeks
  Arms: NGM120 Treatment Group B; NGM120 Treatment Group E

SUMMARY:
A multi-center evaluation of NGM120 in a randomized, double-blind, placebo-controlled study in participants with colorectal cancer who have cancer cachexia.

DETAILED DESCRIPTION:
Evaluation of Efficacy, Safety and Tolerability of NGM120 in a Phase 2, Randomized, Double-blind, Placebo-controlled, Multi-center Study in Participants with Colorectal Cancer who have Cancer Cachexia

ELIGIBILITY:
Inclusion Criteria:

1. Documented active diagnosis of colorectal cancer.
2. Cachexia defined by Fearon criteria of weight loss.
3. Signed informed consent.

Exclusion Criteria:

1. Current active reversible causes of decreased food intake.
2. Receiving tube feedings or parenteral nutrition at the time of Screening or Randomization.
3. Have cachexia caused by other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body weight at Week 12 | 12 Weeks
  To evaluate the effect of NGM120 compared to placebo on body weight.
Treatment-emergent adverse events (TEAEs) characterized by type, frequency, severity, timing, seriousness, and relationship to study drug | 44 Weeks
  To evaluate safety and tolerability of NGM120

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals, Inc
Locations (1):
- NGM Clinical Study Site, Laredo, Texas, United States